CLINICAL TRIAL: NCT00697723
Title: Arterial Versus Venous Graft Recruitment by Intra-Aortic Balloon Pump
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Magna Graecia (Other)
Responsible Party: University of Magna Graecia - Cardiac Surgery Unit
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: UMGIABPrecruit
Record Dates: First submitted 2008-06-11; First posted 2008-06-16 (Estimated); Last update posted 2008-06-16 (Estimated); Status verified 2008-06

CONDITIONS: Coronary Artery Disease
Keywords: Coronary artery bypass graft; Intra-aortic balloon pump; transit-time flowmetry
MeSH Terms: conditions — Coronary Artery Disease

INTERVENTIONS:
Procedure: Transit-time flowmetry — Transit-time flowmetry during 1:1 IABP assistance and when IABP is turned off

SUMMARY:
The aim of this study is to evaluate the different performance of arterial and venous graft with intra-aortic balloon pump support following coronary artery bypass.

ELIGIBILITY:
Inclusion Criteria:

* All patients undergoing coronary artery bypass surgery

Exclusion Criteria:

* Aortic insufficiency;
* Diffuse atherosclerosis impeding intra-aortic balloon pump introduction

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 138 (Actual)
Dates: Start 2005-01; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
Hospital mortality and morbidity | three years

SECONDARY OUTCOMES:
Transit-time flowmetry | three years

CONTACTS AND LOCATIONS:
Locations (1):
- University of Magna Graecia - Cardiac Surgery unit, Catanzaro, Italy

REFERENCES:
- [Result] Baskett RJ, Ghali WA, Maitland A, Hirsch GM. The intraaortic balloon pump in cardiac surgery. Ann Thorac Surg. 2002 Oct;74(4):1276-87. doi: 10.1016/s0003-4975(02)03663-9. PMID 12400798
- [Result] Christenson JT, Simonet F, Badel P, Schmuziger M. Evaluation of preoperative intra-aortic balloon pump support in high risk coronary patients. Eur J Cardiothorac Surg. 1997 Jun;11(6):1097-103; discussion 1104. doi: 10.1016/s1010-7940(97)00087-0. PMID 9237594
- [Result] Tedoriya T, Kawasuji M, Sakakibara N, Takemura H, Watanabe Y, Hetzer R. Coronary bypass flow during use of intraaortic balloon pumping and left ventricular assist device. Ann Thorac Surg. 1998 Aug;66(2):477-81. doi: 10.1016/s0003-4975(98)00468-8. PMID 9725388
- [Result] Yoshitani H, Akasaka T, Kaji S, Kawamoto T, Kume T, Neishi Y, Koyama Y, Yoshida K. Effects of intra-aortic balloon counterpulsation on coronary pressure in patients with stenotic coronary arteries. Am Heart J. 2007 Oct;154(4):725-31. doi: 10.1016/j.ahj.2007.05.019. PMID 17893000